CLINICAL TRIAL: NCT00199719
Title: Study of the Pharmacokinetic Action of Amantadine and Ribavirin in Chronic Hepatitis C Non 2 -3 Genotype naïve Patients Treated With a 12 Weeks Bitherapy of Peginterferon Alpha 2a-ribavirin, and Followed by a Tritherapy of Peginterferon Alpha 2a-ribavirin-amantadine for 36 Weeks
Brief Title: Study of the Pharmacokinetic Action of Amantadine and Ribavirin in Chronic Hepatitis C. CINAM
Acronym: CINAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I02022
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2007-06

CONDITIONS: Chronic Hepatitis C
Keywords: drug monitoring; ribavirin-pharmacokinetic; pharmacodynamics; chronic hepatitis C; non 2 non 3 genotype
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

INTERVENTIONS:
Drug: Ribavirine

SUMMARY:
Peg interferon and ribavirin currently represent the standard approved association for treating patients infected with hepatitis C virus (HCV) . The adjunction of amantadine is expected to gain about 10 % of sustained virological response (SVR) . Unfortunately, about 50 % of the patients remain relapsers or virological non responders. The main predictive factors of SVR are HCV genotype and body weight (BW). The impact of the drug pharmacological properties, particularly those of ribavirin requires complementary studies. This drug has a large distribution volume and its concentrations display large inter-individual variability. Two studies performed in HCV patients found no correlation between ribavirin dose adjusted on BW and a single ribavirin time point serum concentration at steady state.

The aim of this study is to investigate the pharmacokinetic-pharmacodynamic relationships of ribavirin in hepatitis C patient

DETAILED DESCRIPTION:
The study is conducted in naive patients infected with genotype non 2 non 3 administered peginterferon alpha 2-a (40KD) weekly, and ribavirin with dose adjusted on BW (< 75 kg 1000 mg/day, >75 kg 1200 mg/day) for the first three months with adjunction of amantadine 200 mg daily for the following 9 months.

Plasma concentration profiles of ribavirin were studied after the first dose (D0) and at W12. At each period, blood samples were collected pre-dose and 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours post-dosing. Ribavirin concentrations were measured using liquid chromatography-tandem mass spectrometry and ribavirin area under the concentration-timcurves (AUC0-10h) were derived from plasma concentrations profiles using the linear trapezoidal rule.

Virological follow-up was performed at W2, W4, W6, W8, W12, W24 and W72. Early virological response was defined by undetectable viral load at W12.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >18 years of age and <65 years of age
* Génotype non2 non3
* Chronic liver disease consistent with chronic hepatitis C infection on a biopsy (obtained within the past 24 months) as judged by a local pathologist (Metavir >A1and >F1)
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* IFN or ribavirin therapy at any previous time
* Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, anti-HIV Ab
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
-Study of the complete pharmacokinetics of ribavirin at day 1, and day 84 (week 12).
-Study of the complete pharmacokinetics of amantadin and ribavirin at week 12 + one day and at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Véronique LOUSTAUD-RATTI, MD, Principal Investigator — University Hospital, Limoges
Locations (2):
- France (2):
  - Service d'Hépato-gastroentérologie, Angers
  - Service d'Hépatogastroentérologie, Limoges

REFERENCES:
- [Result] Loustaud-Ratti V, Alain S, Rousseau A, Hubert IF, Sauvage FL, Marquet P, Denis F, Lunel F, Cales P, Lefebvre A, Fauchais AL, Liozon E, Vidal E. Ribavirin exposure after the first dose is predictive of sustained virological response in chronic hepatitis C. Hepatology. 2008 May;47(5):1453-61. doi: 10.1002/hep.22217. PMID 18435468